CLINICAL TRIAL: NCT01133496
Title: Open Label, Balanced, Randomized, Two-way, Single-dose, Crossover Bioequivalence Study of Alendronate Sodium 70 mg Tablets of Dr Reddy's, India and Fosamax® Tablets of Merck & Co., Inc., USA, in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Alendronate Sodium Tablets 70 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. Indu Bhushan/Senior Director - R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 095-06
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Alendronate Sodium; crossover
MeSH Terms: interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate Sodium (Experimental): Alendronate Sodium Tablets, 70 mg of Dr. Reddy's
  Interventions: Drug: Alendronate Sodium Tablets, 70 mg
- Fosamax (Active Comparator): Fosamax Tablets 70 mg of Merck & Company. Inc., USA.
  Interventions: Drug: Alendronate Sodium Tablets, 70 mg

INTERVENTIONS:
Drug: Alendronate Sodium Tablets, 70 mg — Alendronate Sodium Tablets, 70 mg of Dr. Reddy's Laboratories Limited.
  Other Names: Fosamax Tablets 70 mg

SUMMARY:
The purpose of this study is to determine the bioequivalence of Alendronate Sodium 70 mg of Dr. Reddy's and Fosamax Tablets 70 mg of Merck & Co.

DETAILED DESCRIPTION:
Open label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover oral bioequivalence study of Alendronate sodium 70 mg tablets of Dr Reddy's Laboratories Limited, India and Fosamax® tablets of Merck & Co., Inc., USA, in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human subjects aged between 18 and 45 years (including both).
2. Subjects with a BMI between 18.5 - 24.9 Kg/m2 but weight not less than 45 Kgs.
3. Female subjects who are postmenopausal or surgically sterile.
4. Female subjects of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD) or abstinence.
5. Subjects with normal health as determined by personal medical history, clinical examination, and laboratory examinations and serology tests.
6. Subjects having normal 12-lead electrocardiogram (ECG).
7. Subjects having normal chest X-Ray (P/A view).
8. Subjects able to communicate effectively.
9. Subjects willing to given written informed consent and adhere to all the requirements of this protocol.

Exclusion Criteria:

1. Subjects having contraindications or hypersensitivity to Alendronate sodium or related drugs.
2. History or presence of any medical condition or disease according the opinion of the physician.
3. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
4. History or presence of significant alcoholism or drug abuse in the past one year.
5. History or presence of significant smoking (more than 10 cigarettes or beedi's/day or consumption of tobacco products).
6. Difficulty with donating blood.
7. Difficulty in swallowing solids like tablets or capsules.
8. Systolic blood pressure less than 90 mm Hg or more than 140 mm Hg.
9. Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
10. Pulse rate less than 50/minute or more than 100/minute.
11. Use of any prescribed medication during last two weeks or OTC medical products during the last one week preceding the first dosing.
12. Major illness during 3 months before screening.
13. Participation in a drug research study within past 3 months.
14. Donation of blood in the past 3 months before screening.
15. Female volunteers demonstrating a positive pregnancy screen.
16. Female volunteers who are currently breast-feeding.
17. Female volunteers with child bearing potential using prohibited contraceptive method (Oral, Injectable or Implantable hormonal agents).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Naba Kr Talukdar, MD, Principal Investigator — GVK Biosciences Pvt. Ltd.
Locations (1):
- GVK Biosciences Pvt. Ltd.,, Hyderabad, Andhra Pradesh, India